CLINICAL TRIAL: NCT00667771
Title: Effect of Naltrexone on Craving and Ethanol-Induced Brain Activity
Brief Title: The Effect of Naltrexone on Alcohol Craving and on Brain Activity During Alcohol Infusion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 080125; 08-AA-0125
Record Dates: First submitted 2008-04-25; First posted 2008-04-28 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-04

CONDITIONS: Alcohol Dependence; Alcoholism
Keywords: Alcohol; Naltrexone; fMRI; Alcoholism; Alcoholics; Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

INTERVENTIONS:
Drug: Naltrexone

SUMMARY:
This study will determine whether naltrexone, a medicine used to treat alcoholism, can lessen the craving for alcohol during alcohol withdrawal and examine how the drug affects brain activity during alcohol infusion.

People between 21 and 50 years of age who are right-handed, alcohol-dependent, and have at least one family member with a history of alcoholism, may be eligible for this study.

Participants are admitted to the NIH Clinical Center for 1 month for the following procedures:

Screening

* Medical history, alcohol-use history and family history of alcoholism
* Physical examination, psychological tests and blood tests
* Medicine to lessen alcohol withdrawal symptoms, if necessary

Days 1-7

* Alcohol detoxification
* Medical and psychological evaluations
* Assignment to naltrexone or placebo group

Days 7 through 28

* Drug treatment: Take naltrexone or placebo capsule every morning
* Additional alcohol-dependence treatment: Cognitive and behavioral therapies and participation in self-help groups, such as Alcoholics Anonymous
* Weekly questionnaires to measure mood and desire for alcohol
* Blood tests
* Alcohol craving stimulation test (day 7): Subjects handle and sniff water and then their favorite alcoholic beverage. They then rate their urge to drink alcohol and their level of anxiety and their heart rate is measured.
* Alcohol infusion test (day 9): Subjects have an MRI scan during infusion through a vein of saline (salt water), followed by infusion of alcohol. For this test, a catheter (plastic tube) is placed in a vein in each arm, one for administering the saline and then alcohol; the other for drawing blood samples to measure blood alcohol level and body chemistries. Before, during and after the infusion, subjects are asked to respond to questions about their feelings, cravings and mood changes.

Follow-up

Subjects are asked to participate in a 3-month outpatient assessment program involving five outpatient visits (at 1, 2, 4, 8 and 12 weeks after discharge). At each visit, they fill out questionnaires and to take a breathalyzer test and blood and urine tests for drugs. They may continue naltrexone therapy and weekly group therapy sessions during this time. Subjects who do not participate in the assessment program are contacted at home by phone once a week for 1 month and then every other week for the next 2 months to monitor alcohol abstinence.

...

DETAILED DESCRIPTION:
Alcoholism is a chronic, progressive, brain disorder with a profound impact on individuals' lives and economic cost to society. The positive reinforcing effect of alcohol is a key element in the transitional development from alcohol intake to alcohol addiction. Findings from animal and human studies indicate that the rewarding properties of ethanol arise in part from a complex interaction between alcohol, endogenous opioids, and dopamine (DA) systems. Acute administration of ethanol increases the release of opioid peptides, which in turn, increases the release of DA in the mesocorticolimbic system. Naltrexone (NTX), an opioid receptor antagonist, has been studied widely in both preclinical and clinical research for the treatment of alcoholism. Numerous clinical studies have shown that short-term use of NTX on alcohol-dependent patients effectively prevents relapse and reduces the level of craving. Genetic studies have suggested that individuals with mu-opioid receptors (OPRMs) encoded by the 118G gain-of function variant allele experience a greater therapeutic response to NTX. There are no data utilizing functional Magnetic Resonance Imaging (fMRI) to study the effect of NTX on brain activity during an intravenous (IV) infusion of ethanol.

Objectives:

To study the effect of NTX on the blood oxygen level dependent (BOLD) response in the ventral striatum area of the brain in response to an ethanol infusion.

To study the effect of NTX on cue reactivity (CR) to alcohol-associated cues.

Study population:

Alcohol-dependent patients between the ages of 21-50 years.

Design:

All participants will complete a screening telephone interview before coming to the NIAAA Inpatient Unit. The interviewer will inform eligible participants about the requirements and procedures associated with current protocols. Following admission to NIAAA Inpatient Unit, all participants will be enrolled in the Assessment and Treatment of People with Alcohol Drinking Problems protocol (#05-AA-0121). Protocol 05-AA-0121 will allow us to evaluate each participant's general medical and psychiatric conditions and provide standard of care for treatment seeking alcoholics.

Participants, who fulfill the specific requirements of the NTX protocol, will be thoroughly informed about the nature of the study before obtaining an informed consent. Consented participants will be randomized, using a double-blind design, to receive either 50 mg of NTX per day or placebo. Medications will be administered at 8:00 AM on a daily basis by the nursing staff.

Prior to the challenge procedures (CR on Day 7 and fMRI/ethanol infusion on Day 9), a clinical nurse specialist who is not involved with the protocol will re-consent each participant when they are not in acute withdrawal. The re-consenting process will provide reassurance that participants understand the requirements and implications associated with participation in the CR and fMRI/ethanol infusion procedures. Individuals who elect not to participate in the CR and fMRI/ethanol infusion sessions will be discharged from the in-patient unit and encouraged to continue treatment in the NIAAA Outpatient Clinic for the next three months.

Participants who elect to remain in the study will take part in the CR session on Day 7 and fMRI/ethanol infusion session on Day 9 (procedures are described on Page 13 under study procedures). Following the fMRI/ethanol infusion session, participants will remain in the hospital for approximately three weeks to monitor their craving and take part in our inpatient treatment program for alcoholism. During the post-challenge hospitalization, all participants will be offered 50 mg of NTX once a day. Following discharge from the hospital, participants will be encouraged to continue treatment in NIAAA Outpatient Clinic for three months.

Outcome Measures:

BOLD response during the ethanol infusion challenge.

BOLD brain response to emotional facial stimuli.

Self-reported Alcohol Urge Questionnaires (AUQ), Penn Alcohol Craving Scale (PACS), Obsessive Compulsive Drinking Scale (OCDS) and Profile of Mood Status (POMS).

Hormonal responses to the ethanol challenge: plasma ACTH, cortisol, and beta-endorphin.

Subjective responses to the ethanol challenge as rated by stimulation, sedation, high, and intoxication questionnaires.

Cue-induced craving during the CR session.

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants must:

* be right-handed
* between 21 and 50 years of age
* meet the DSM-IV diagnostic criteria for alcohol dependence (polysubstance abuse is common in younger alcohol-dependent patients, and will not be exclusionary)
* have a positive family history of alcoholism (one or more first-degree relatives with alcohol problems)

In addition, female participants:

* must have a negative urine pregnancy test (beta-hCG)
* of childbearing capability will be required to use a double contraceptive method (such as oral contraceptives, condom with spermicide or intra-uterine device with spermicide) from the start of the study until at least one month following the last dose of NTX.

EXCLUSION CRITERIA:

General exclusion criteria for the NIAAA Intramural treatment program:

* people who present with complicated medical problems requiring intensive medical or diagnostic management, such as uncontrolled hypertension, gastro-intestinal (GI) bleeding, major organ or body system dysfunction or thyroid disease
* people who are infected with human immunodeficiency virus (HIV)
* serious neuro-psychiatric conditions which impair judgment or cognitive function to an extent that precludes them from providing informed consent or complying with study procedures, such as psychotic illness, or severe dementia (individuals not competent to give informed consent)
* people who are unlikely or unable to complete the study because they are likely to be incarcerated while on the protocol
* people who are required to receive treatment by a court of law or who are involuntarily committed to treatment

Specific exclusion criteria for this protocol include:

* clinically significant hepatobiliary disease
* a history of facial flushing in response to alcohol
* a history of seizures
* currently psychotic
* currently abusing opioids
* use of psychotropic medications (antidepressant, lithium, antipsychotic, anxiolytic, antiepileptic) regularly within the last 4 weeks prior to admission
* having a positive pregnancy test, contemplating pregnancy in the next 3 months, nursing, or not using an effective contraceptive method (if the participant is of child-bearing potential)
* a history of allergy or unusual reactions to NTX
* have received treatment with NTX in the six-month period prior to enrollment
* presence of ferromagnetic brain aneurysm clips, implanted pacemaker, hearing aid, or any other metallic implant, such as pins, screws, plates, dentures, or non-removable jewelry, in or on the body
* pronounced claustrophobia

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2008-04-22; Primary Completion 2010-12-27 (Actual); Study Completion 2011-04-04 (Actual)

PRIMARY OUTCOMES:
BOLD response during the ethanol infusion challenge

SECONDARY OUTCOMES:
Self-reported AUQ, PACS, OCDS, POMS and cue-induced craving during the CR session

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Appel SB, Wise L, McDaid J, Koyama S, McElvain MA, Brodie MS. The effects of long chain-length n-alcohols on the firing frequency of dopaminergic neurons of the ventral tegmental area. J Pharmacol Exp Ther. 2006 Sep;318(3):1137-45. doi: 10.1124/jpet.106.105148. Epub 2006 Jun 1. PMID 16740620
- [Background] Barr CS, Schwandt M, Lindell SG, Chen SA, Goldman D, Suomi SJ, Higley JD, Heilig M. Association of a functional polymorphism in the mu-opioid receptor gene with alcohol response and consumption in male rhesus macaques. Arch Gen Psychiatry. 2007 Mar;64(3):369-76. doi: 10.1001/archpsyc.64.3.369. PMID 17339526
- [Background] Bart G, Kreek MJ, Ott J, LaForge KS, Proudnikov D, Pollak L, Heilig M. Increased attributable risk related to a functional mu-opioid receptor gene polymorphism in association with alcohol dependence in central Sweden. Neuropsychopharmacology. 2005 Feb;30(2):417-22. doi: 10.1038/sj.npp.1300598. PMID 15525999
- [Derived] Spagnolo PA, Ramchandani VA, Schwandt ML, Zhang L, Blaine SK, Usala JM, Diamond KA, Phillips MJ, George DT, Momenan R, Heilig M. Effects of naltrexone on neural and subjective response to alcohol in treatment-seeking alcohol-dependent patients. Alcohol Clin Exp Res. 2014 Dec;38(12):3024-32. doi: 10.1111/acer.12581. PMID 25581657